CLINICAL TRIAL: NCT05970172
Title: A Phase 3, Open-label, Uncontrolled Study to Evaluate the Activity, Safety, Pharmacokinetics and Pharmacodynamics of Roxadustat for the Treatment of Anemia in Pediatric Participants With Chronic Kidney Disease
Brief Title: A Study of Roxadustat to Treat Anemia in Children and Teenagers With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-1003; 2022-501980-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-07-25; First posted 2023-08-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Renal Anemia
Keywords: Roxadustat; ASP1517; Pediatric; Renal Anemia; Chronic renal failure; Chronic Kidney Disease; Renal Insufficiency, Chronic; Anemia; Open-label; Uncontrolled; Safety; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Roxadustat (Experimental): Participants will receive roxadustat orally (or via gastric tube as an aqueous dispersion, if necessary) 3 times per week. The 24-week treatment period is defined as 4 weeks of fixed dose treatment followed by 20 weeks of dose titration(s). Dose titrations will be based on hemoglobin (Hb) monitoring. Participants in the study may receive roxadustat treatment for up to 52 weeks.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Oral
  Other Names: ASP1517; FG-4592; Evrenzo

SUMMARY:
Roxadustat is a licensed medicine to treat anemia in adults with chronic kidney disease (CKD). Anemia is a low level of red blood cells. Current treatment for anemia is to have injections of medicines called erythropoietin stimulating agents (also known as ESAs) to help the bone marrow make more red blood cells. These are often given together with iron. This treatment is also available to children and teenagers with CKD. However, there are some safety concerns with ESAs. Also, as roxadustat is taken orally, this may be another option for treating anemia in children and teenagers with CKD. In this study, children and teenagers with CKD and anemia will take roxadustat for up to 52 weeks to treat their anemia.

The main aim of the study is to learn how roxadustat affects anemia in children and teenagers with CKD.

This is an open-label study which means the children and teenagers in the study and the clinic staff know they will be taking roxadustat. In this study, the children and teenagers with CKD who need treatment for anemia can take part. Those currently being treated with an ESA will be switched to roxadustat. Those who have not been treated with an ESA can start on roxadustat straight away. All children and teenagers in the study will take roxadustat 3 times a week for up to 52 weeks (1 year). They will start on a fixed dose of roxadustat for 4 weeks. Blood samples will be taken regularly to check hemoglobin levels. The roxadustat dose may be changed if the blood levels of hemoglobin are too high, too low, or change too quickly. After 4 weeks the dose may be changed, if needed, to keep blood levels of hemoglobin in the blood to just below the normal range.

Firstly, teenagers will take roxadustat. 10 teenagers will take their fixed dose of roxadustat for 4 weeks. They will give blood samples to help the researchers work out the most suitable dose for the rest of the teenagers in the study. When the rest of the teenagers start taking roxadustat at the most suitable dose for teenagers, 10 children will take roxadustat for 4 weeks. These 10 children will give blood samples to help the researchers work out the most suitable dose for the rest of the children in the study. Then, the rest of the children will take roxadustat at the most suitable dose for children.

There will be many clinic visits during the study. Overnight hospital stays are not expected. There will be 1 visit every 2 weeks for the first 4 weeks of taking roxadustat, then every 4 weeks until the end of treatment. Finally there is 1 visit 4 weeks after treatment has finished.

During most visits, the children and teenagers will have their vital signs checked (blood pressure, body temperature and heart rate). Fluid status (how much water is in the body) will also be checked for those who need dialysis. The children and teenagers will also have blood tests and the study doctors will check for any medical problems. The children and teenagers will have a medical examination before their first dose of roxadustat and again at about 24-week (6-month) and 52-week (13-month) visits. They will have an electrocardiogram (ECG) before their first dose of roxadustat and again at the 12-week, 24-week, 36-week, and 52-week visit. They will also have urine tests at the 4-week, 24-week and 52-week visits. At the 52-week visit, the children and teenagers will also have blood tests for hemoglobin and iron levels. The study doctors will also check for any medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of anemia in CKD Kidney Disease Outcomes Quality Initiative stages 3 or 4 or 5. This can include participants not on dialysis or dialysis dependent (DD) participants (including hemodialysis, peritoneal dialysis and hemodiafiltration participants).
* Participants not on dialysis must have an estimated glomerular filtration rate (Schwartz formula) of < 60 mL/min per 1.73 m^2.
* ESA-treated participants should have a screening Hb level, assessed via HemoCue, between 10.0 and 12.0 g/dL; ESA-naïve participants can have a Hb level ≤ 11 g/dL.
* Participant has a ferritin level > 100 ng/mL or a transferrin saturation (TSAT) value > 20%.
* Participant has an alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 x upper limit of normal (ULN) and total bilirubin (TBL) ≤ 1.5 x ULN at enrollment visit.
* Participant is treated with an ESA or is ESA-naïve, where ESA status is defined as:

  * ESA-treated: Participant is taking a stable dose of an ESA for at least 4 weeks prior to screening.
  * ESA-naïve: Participant has no prior ESA exposure OR participant's total prior ESA exposure ≤ 3 weeks within the preceding 4 weeks from screening OR participant was previously treated with and discontinued an ESA ≥ 8 weeks prior to screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 4 weeks after final study intervention administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study and for 4 weeks post-last roxadustat dose.
* Female participant must not donate ova starting at first administration of roxadustat and throughout the study period and for 4 weeks post-last roxadustat dose.
* Male participants with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 4 weeks post-last roxadustat dose.
* Male participants must not donate sperm during the treatment period and for 4 weeks post-last roxadustat dose.
* Male participants with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 4 weeks post-last roxadustat dose.
* Participant and/or participant's parent or legal guardian agrees for the participant not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any medical condition, including active, systemic or clinically significant infection which may pose a safety risk to a participant in this study, which may confound the safety or activity assessment or may interfere with study participation making the participant unsuitable for study.
* Participant has a known or suspected hypersensitivity to roxadustat, related hypoxia-inducible factor-prolyl hydroxylase inhibitors (HIF-PHI), or any components of the formulation used.
* Participant has uncontrolled hypertension (defined as ≥ 95th percentile + 12 mm Hg or ≥ 140/90 mm Hg [whichever is lower] for participants < 13 years of age and ≥ 140/90 mm Hg for participants ≥ 13 years of age measured 3 times at the same visit) in the 2 weeks prior to screening.
* Participant has a known hematologic disease other than anemia secondary to renal disease,(e.g., history of sickle cell disease, sickle cell anemia, hemoglobin sickle cell disease, or hemoglobin sickle cell beta thalassemia).
* Participant has untreated hypothyroidism.
* Participant has severe hyperparathyroidism defined as serum parathyroid hormone (PTH) levels above 1000 pg/mL intact PTH within 4 weeks of screening.
* Participant has a functioning kidney allograft.
* Participant has a folate or B12 or carnitine deficiency. Acceptable if treated to normal values within 4 weeks of screening.
* Participant has a known active malignancy or malignancy within 18 months before the screening visit. Radiation or chemotherapy must be completed at least 12 months before the screening visit.
* Participant has a scheduled living donor organ transplantation date within 12 weeks of screening. If participant becomes eligible for a kidney transplant during study conduct, the participant should be discontinued.
* Participant has a whole blood or packed red blood cells (pRBC) transfusion during the 8 weeks prior to screening.
* Participant has any current condition leading to active significant blood loss in the past 4 weeks.
* Participant has a diagnosis of hemolytic uremic syndrome within 12 weeks prior to screening.

  * Participant who has a previous diagnosis of atypical hemolytic syndrome must be relapse-free (stable hemoglobin (Hb), normal platelet count, normal serum lactate dehydrogenase, and normal haptoglobin level) for more than 12 weeks prior to screening.
* Participant has a history of chronic liver disease, including comorbidity with autosomal recessive polycystic kidney disease, cystinosis, and primary hyperoxaluria.
* Participant had an episode of peritonitis within 30 days of screening.
* Participant has active inflammation such as glomerulonephritis flare (i.e., lupus nephritis, immunoglobulin A (IgA) nephritis, rapidly progressive glomerulonephritis, membranoproliferative glomerulonephritis, antineutrophil cytoplasmic antibodies vasculitis) requiring pulse corticosteroid treatment or induction treatment with an immunosuppressive agent (i.e., cyclophosphamide, rituximab, or another monoclonal antibody) within 6 weeks of screening visit. Receipt of monoclonal antibody or biologic for maintenance treatment of underlying condition is acceptable.
* Participant has a known history of human immunodeficiency virus infection.
* Participant has rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption or is allergic to peanut or soya.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hb level to the average Hb level over treatment weeks 20 to 24 | Baseline and weeks 20 to 24
  Mean change in Hb level between baseline and average Hb level over treatment weeks 20 to 24.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of roxadustat in plasma: Maximum concentration (Cmax) | Up to week 8
  Cmax will be recorded from the PK plasma samples collected.
PK of roxadustat in plasma: Area under the plasma-concentration time curve (AUC) | Up to week 8
  AUC will be recorded from the PK plasma samples collected.
PK of roxadustat in plasma: Apparent total clearance (CL/F) | Up to week 8
  CL/F will be recorded from the PK plasma samples collected.
PK of roxadustat in plasma: Time of the maximum concentration (Tmax) | Up to week 8
  Tmax will be recorded from the PK plasma samples collected.
Hb levels at all timepoints | Up to week 56
  Hb levels at all timepoints will be recorded.
Dose titration history at all timepoints | Up to week 52
  Dose titration history at all timepoints will be recorded.
Number of participants with treatment-emergent adverse events (TEAEs) | From first dose of study drug and up to week 56
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of roxadustat, whether or not considered related to roxadustat. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of roxadustat. This includes events related to the comparator and events related to the (study) procedures. A TEAE is defined as an AE observed after starting administration of roxadustat through 28 days after the last dose of roxadustat.
Number of participants with treatment-emergent cardiovascular AEs | From first dose of study drug and up to week 56
  Treatment-emergent cardiovascular AEs will be recorded.
Number of participants with treatment-emergent thrombotic AEs | From first dose of study drug and up to week 56
  Treatment-emergent thrombotic AEs will be recorded.
Number of participants with laboratory value abnormalities and/or AEs | Up to week 52
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to week 52
  Number of participants with potentially clinically significant vital sign values.
Change from baseline in growth parameter value: Height | Baseline and up to week 52
  Height will be recorded at all timepoints.
Change from baseline in growth parameter value: Weight | Baseline and up to week 52
  Weight will be recorded at all timepoints.
Number of participants with physical examinations abnormalities and/or AEs | Up to week 52
  Number of participants with potentially clinically significant physical examination abnormalities.
Percentage of participants with Hb response | Up to Week 24
  Response is defined as a participant achieving 2 consecutive Hb values within 1 g/dL of baseline (ESA-treated participants only) or achieving the target range of 10.0 to 12.0 g/dL at the end of the 24-week treatment evaluation period (i.e., weeks 20 to 24) without having received rescue therapy within 6 weeks prior to or during this 4-week evaluation period.
Mean monthly intravenous (IV) iron use | Up to week 52
  Summaries of monthly IV iron usage (number of administrations) will be recorded.
Mean Monthly total IV iron dosage | Up to week 52
  Summaries of monthly IV iron usage (total dosage) will be recorded.
Percentage of participants using IV iron | Up to week 52
  Percentage of participants using IV iron by study period will be recorded.
Percentage of participants using oral iron | Up to week 52
  Percentage of participants using oral iron by study period will be recorded.
Percentage of participants using rescue therapy | Up to week 52
  Percentage of participants using rescue therapy by study period will be recorded.
Palatability questionnaire | Up to week 52
  The palatability questionnaire will assess taste and ability to swallow the medication using a 5 point Likert scale: for taste from 0 (Really bad) to 4 (Really good); for ability to swallow from 0 (Really Difficult) to 4 (Really Easy). The number of participants recorded for each response category will be provided.
Change from baseline in Pediatric Quality of Life (PedsQL) Inventory Score | Baseline and up to week 52
  PedsQL Inventory Scale comprises of 23 items (except for ages 2-4 which has only 21 items, 3 of which are only answered if the child attends school or daycare) in 4 domains: physical functioning, emotional functioning, social functioning and school functioning. A Likert scale from 0 (Never) to 4 (Almost always) will be used to record response. Higher scores indicate better quality of life.
Change from baseline in PedsQL Multidimensional Fatigue Scale questionnaire QoL Score | Baseline and up to week 52
  PedsQL Multidimensional Fatigue Scale comprises of 18 items in 3 domains: general fatigue, sleep/rest fatigue and cognitive fatigue. A Likert scale from 0 (Never) to 4 (Almost always) will be used to record response. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (46):
- Belgium (4):
  - Site BE32002, Brussels
  - Site BE32001, Edegem
  - Site BE32004, Ghent
  - Site BE32003, Leuven
- Site BG35901, Sofia, Bulgaria
- Croatia (2):
  - Site HR38501, Zagreb
  - Site HR38503, Zagreb
- Czechia (2):
  - Site CZ42002, Brno
  - Site CZ42001, Prague
- Site DK45001, Aarhus, Denmark
- Site DE49001, Tübingen, Germany
- Greece (2):
  - Site GR30002, Athens
  - Site GR30001, Thessaloniki
- Site IE35301, Dublin, Ireland
- Italy (2):
  - Site IT39003, Milan
  - Site IT39004, Padua
- Site LB96101, El Achrafiyé, Lebanon
- Site LT37001, Vilnius, Lithuania
- Site NL31002, Rotterdam, Netherlands
- Site NO47002, Oslo, Norway
- Poland (2):
  - Site PL48003, Krakow
  - Site PL48002, Warsaw
- Romania (2):
  - Site RO40002, Clug Napoca
  - Site RO40001, Timișoara
- Saudi Arabia (2):
  - Site SA96602, Dammam
  - Site SA96601, Riyadh
- Site SK42101, Bratislava, Slovakia
- Spain (2):
  - Site ES34003, Esplugues de Llobregat
  - Site SP34001, Madrid
- Sweden (2):
  - Site SE46002, Mölnlycke
  - Site SE46003, Mölnlycke
- Turkey (Türkiye) (8):
  - Site TR90001, Ankara
  - Site TR90007, Ankara
  - Site TR90010, Ankara
  - Site TR90003, Istanbul
  - Site TR90008, Istanbul
  - Site TR90005, İzmit
  - Site TR90006, Kayseri
  - Site TR90002, Manisa
- United Kingdom (7):
  - Site GB44005, Cardiff
  - Site GB44006, Glasgow
  - Site GB44008, Liverpool
  - Site GB44007, London
  - Site GB44003, Newcastle upon Tyne
  - Site GB44001, Nottingham
  - Site GB44004, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/